CLINICAL TRIAL: NCT00220792
Title: A Multicenter Trial of Group Therapy for Breast Cancer
Brief Title: Group Therapy for Primary Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cummings Foundation (Unknown)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CA61309
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Primary breast cancer; support groups; mood disturbance
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Behavioral: Brief supportive-expressive group therapy

SUMMARY:
The purpose of this study is to determine whether women with primary breast cancer who were randomly assigned to receive a brief group therapy would show a greater reduction in mood disturbance over time compared to those randomized to the control condition. We also hypothesized that women who were highly distressed at baseline would show the greatest benefit from participating in a support group, and that therapists with more training and experience would be most effective in reducing distress.

DETAILED DESCRIPTION:
Breast cancer patients often experience significant psychological distress after diagnosis and during initial treatment. Group interventions for cancer patients have been shown to improve psychological adjustment. The tests of efficacy for these interventions have typically taken place in university settings using highly developed models of intervention. Our aim was to test our supportive-expressive model in community oncology practices utilizing personnel already working with these populations. To conduct this study of group therapy for primary breast cancer patients, we developed a brief version of the supportive-expressive model (Classen et al., 1993). Our first aim was to test the efficacy of this intervention for reducing mood disturbance for women who received the intervention compared to a control group. A second aim was to examine who was most likely to benefit from the intervention. A third aim was to see if this method could be taught efficiently and effectively to oncology nurses and mental health professionals.

ELIGIBILITY:
Inclusion Criteria:

* : 1) diagnosis of primary, biopsy-proven breast cancer, stages I through IIIA; 2) diagnosis occurred no more than 12 months prior to recruitment; 3) completion of initial surgical treatment; and 4) no detectable disease present.

Exclusion Criteria:

* 1) evidence of metastases beyond adjacent lymph nodes, including chest wall involvement, bone or viscera; 2) recurrence of the cancer prior to randomization; 3) diagnosis of other cancers (except for basal cell or squamous cell carcinoma of the skin or in situ cervical cancer) within the past 10 years; 4) any other major medical problems likely to limit life expectancy to less than 10 years; 5) a history of major psychiatric illness for which the patient was hospitalized or medicated, except for a diagnosis of depression or anxiety treated for a period of less than one year; and 6) attendance at a cancer support group for more than two months.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480
Dates: Start 1993-06; Study Completion 1998-06

PRIMARY OUTCOMES:
Rate of change in mood disturbance assessed by the Profile of Mood States at baseline, 3 mo, 6 mo, 12 mo, 18 mo and 24 mo.

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, MD, Principal Investigator — Stanford University
Locations (10):
- United States (10):
  - Social Work Consultants, Inc, Wichita, Kansas
  - Kalamazoo Community Clinical Oncology Program, Kalamazoo, Michigan
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Northern New Jersey CCOP, Hackensack, New Jersey
  - North Shore University Hospital CCOP, Manhasset, New York
  - University of Rochester CCOP, Rochester, New York
  - Syracuse Hem/Onc CCOP, Syracuse, New York
  - Northwest CCOP, Tacoma, Washington
  - Marshfield Medical Research Foundation, Marshfield, Wisconsin
  - Milwaukee CCOP, Milwaukee, Wisconsin

REFERENCES:
- [Background] Han WT, Collie K, Koopman C, Azarow J, Classen C, Morrow GR, Michel B, Brennan-O'Neill E, Spiegel D. Breast cancer and problems with medical interactions: relationships with traumatic stress, emotional self-efficacy, and social support. Psychooncology. 2005 Apr;14(4):318-30. doi: 10.1002/pon.852. PMID 15386762
- [Background] Fobair P, Koopman C, DiMiceli S, O'Hanlan K, Butler LD, Classen C, Drooker N, Davids HR, Loulan J, Wallsten D, Spiegel D. Psychosocial intervention for lesbians with primary breast cancer. Psychooncology. 2002 Sep-Oct;11(5):427-38. doi: 10.1002/pon.624. PMID 12228876
- [Background] Koopman C, Butler LD, Classen C, Giese-Davis J, Morrow GR, Westendorf J, Banerjee T, Spiegel D. Traumatic stress symptoms among women with recently diagnosed primary breast cancer. J Trauma Stress. 2002 Aug;15(4):277-87. doi: 10.1023/A:1016295610660. PMID 12224799
- [Background] Fobair P, O'Hanlan K, Koopman C, Classen C, Dimiceli S, Drooker N, Warner D, Davids H, Loulan J, Wallsten D, Goffinet D, Morrow G, Spiegel D. Comparison of lesbian and heterosexual women's response to newly diagnosed breast cancer. Psychooncology. 2001 Jan-Feb;10(1):40-51. doi: 10.1002/1099-1611(200101/02)10:13.0.co;2-s. PMID 11180576
- [Background] Spiegel D, Morrow GR, Classen C, Raubertas R, Stott PB, Mudaliar N, Pierce HI, Flynn PJ, Heard L, Riggs G. Group psychotherapy for recently diagnosed breast cancer patients: a multicenter feasibility study. Psychooncology. 1999 Nov-Dec;8(6):482-93. doi: 10.1002/(sici)1099-1611(199911/12)8:63.0.co;2-w. PMID 10607981
- [Background] Classen C, Abramson S, Angell K, Atkinson A, Desch C, Vinciguerra VP, Rosenbluth RJ, Kirshner JJ, Hart R, Morrow G, Spiegel D. Effectiveness of a training program for enhancing therapists' understanding of the supportive-expressive treatment model for breast cancer groups. J Psychother Pract Res. 1997 Summer;6(3):211-8. PMID 9185066
- [Background] Spiegel, D., Morrow, G.R., Classen, C., Riggs, G., Stott, P.B., Mudaliar, N., Pierce, H.I., Flynn, P.J., & Heard, L. (1996). Effects of group therapy on women with primary breast cancer. The Breast Journal, 2(1), 104-106.
- [Background] Azarow, J., Han W.T., Koopman, C., Classen C., Morrow G.R., & Spiegel, D. (2001) Traumatic stress, pain, and self-efficacy are related to breast cancer patients' satisfaction with care. Psychosomatic Medicine, 63, 1, 1130